CLINICAL TRIAL: NCT04003805
Title: Biomarkers of Exposure and Effect in Standardized Research E-cigarette (SREC) Users
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018NTLS016; U01DA045523 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-07-01 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Smoking, Cigarette
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Switching from Smoking Cigarettes to SREC (Experimental)
  Interventions: Drug: Standardized Research E-cigarette (SREC)

INTERVENTIONS:
Drug: Standardized Research E-cigarette (SREC) — The device operates at a single output voltage (3.30 ± 0.05 V) and uses sealed disposable 3-mL cartridges with tobacco-flavored e-liquid (~350 puffs/cartridge). The concentration of nicotine in e-liquid is 15 mg/mL, and the vehicle composition is 50:50 propylene glycol and glycerin. The device uses a battery that can be recharged via a micro USB port. A single charge is designed to sustain more than 400 puffs, which is more than the capacity of an e-liquid cartridge. The e-liquid and the aerosol are well-characterized in terms of chemical impurities and by-products (such as aldehydes), which are minimal. Additional information, including the results of pharmacokinetics study is available via NIDA website: https://www.drugabuse.gov/funding/supplemental-information-nida-e-cig

SUMMARY:
This study is focused on characterizing the toxic and carcinogenic potential of the Standardized Research E-cigarette (SREC) developed by the National Institute on Drug Abuse. In the environment of continuously changing e-cigarette market, SREC was developed as a model e-cigarette that will remain available for an extended period of time and can be used as a bridging element in various studies aimed at evaluating the value and limitations of e-cigarettes as tobacco risk reduction tools. Our overall goal is to generate initial reference data on chemical exposures and associated effects in smokers switching to SREC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female smokers who are 18-65 years of age and are willing to stop smoking and completely switch to e-cigarettes or medicinal nicotine;
* Report smoking ≥ 5 cigarettes daily and not using any other nicotine or tobacco product;
* Biochemically confirmed regular smoking status by a NicAlert test level of 6;
* Smoking daily for at least 1 year and no serious quit attempts (e.g., quit for 24 hours or longer) in the last 3 months (to ensure stability of daily smoking, particularly for those randomized to the continued smoking group);
* No unstable and significant medical or psychiatric conditions as determined by medical history and Prime-MD (to ensure safety of the subject, to minimize the effects of poor health on biomarker measures and to maximize compliance to study procedures);
* Subjects are in good physical health (no unstable medical condition);
* Subjects are in stable, good mental health (e.g. not currently, within the past 6 months, experiencing unstable or untreated psychiatric diagnosis, including substance abuse);
* Subjects who are not taking anti-inflammatory medications or any medications that affect relevant metabolic enzymes;
* Women who are not pregnant or nursing or planning to become pregnant;
* Subject has provided written informed consent to participate in the study (adolescents under the age of 18 will be excluded because this project involves continued use of tobacco products and new tobacco products).

Exclusion Criteria:

* Regular tobacco or nicotine product use (e.g., 9 days in last 30 days) other than cigarettes;
* Currently using nicotine replacement or other tobacco cessation products;
* Significant immune system disorders, respiratory diseases, kidney or liver diseases or any other medical disorders that may affect biomarker data;
* Unstable health conditions (any significant serious, unstable medical condition including, but not limited to, cardiovascular disease, unstable COPD, seizure disorder and cancer, as determined by the licensed medical professional);
* Unstable mental health (to be determined by medical history, CESD, Prime-MD after review by the licensed medical professional);
* Excessive drinking (e.g., 5 or more drinks daily) or problems with drinking or drugs (e.g., self-report of binge drinking alcohol or treatment for drug or alcohol abuse within last 3 months); to be assessed by PI or licensed medical professional;
* Blood alcohol test > 0.01 (g/dL) as measured by a breath sample at screening (participants failing the breath alcohol screen will be allowed to re-screen once;
* Positive toxicology screen for any of the following drugs: cocaine, opiates, methadone, benzodiazepines, barbiturates, amphetamines, methamphetamines, and PCP. Failing temperature strip for the sample. Marijuana will be tested for, but will not be an exclusionary criterion. Participants with valid prescriptions for opiates, benzodiazepines, barbiturates, amphetamines or methadone will not be excluded. Participants failing the toxicology screen will be allowed to re-screen once;
* Pregnant or breastfeeding;
* Failure to agree to take adequate protection to avoid becoming pregnant during the study;
* Vital signs outside of the following range (participants failing for vital signs will be allowed to re-screen once):

  * Systolic BP greater than or equal to 160 mm/hg
  * Diastolic BP greater than or equal to 100 mm/hg
  * Systolic BP below 90 mm/hg and symptomatic (dizziness, extreme fatigue, difficulty thinking, inability to stand or walk, feeling faint)
  * Diastolic BP below 50 mm/hg and symptomatic (dizziness, extreme fatigue, difficulty thinking, inability to stand or walk, feeling faint)
  * Heart rate greater than or equal to 105 bpm
  * Heart rate lower than 45 bpm and symptomatic (dizziness, extreme fatigue, difficulty thinking, inability to stand or walk, feeling faint)
* Expired air carbon monoxide (CO) level greater than 80 ppm;
* Self-reported allergies to propylene glycol or vegetable glycerin;
* Adverse reactions when previously using electronic cigarettes;
* Household member enrolled in the study concurrently;
* Unable to read for comprehension or completion of study documents;
* Unstable living environment that would compromise the ability to attend visits, sequester study products or complete study procedures outside of visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2026-05-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Stepanov, PhD, Principal Investigator — University of Minnesota, Division of Environmental Health Sciences
Locations (1):
- University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Switching From Smoking Cigarettes to SREC: Standardized Research E-cigarette (SREC): The device operates using a rechargeable 400 mAh lithium-ion battery and uses sealed disposable 1.9-mL pods with e-liquid containing 5% w/w nicotine. Flavors that will be available include tobacco, menthol, watermelon and blueberry. The device uses a battery that can be recharged via a micro USB port. The e-liquid and the aerosol are well-characterized in terms of chemical impurities and by-products (such as aldehydes), which are minimal.
Period: Overall Study
Arm/Group | Switching From Smoking Cigarettes to SREC
Started | 47
Completed | 23
Not Completed | 24
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 11
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Switching From Smoking Cigarettes to SREC
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 43
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Exposure Biomarkers: Cotinine
Description: Cotinine (biomarker of nicotine) level after switching to SREC as percentage of baseline level
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of baseline level
Groups:
- Switching From Smoking Cigarettes to SREC: Participants who smoked at baseline were asked to completely switch to SREC e-cigarette for 6 weeks.
Arm/Group | Switching From Smoking Cigarettes to SREC
Number analyzed (Participants) | 23
Percentage of baseline level | 98.5 (51.1)

2. Primary Outcome: Exposure Biomarkers: NNAL
Description: Total NNAL level after switching to SREC as percentage of baseline level
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of baseline level
Arm/Group | Switching From Smoking Cigarettes to SREC
Number analyzed (Participants) | 23
Percentage of baseline level | 53.7 (40.8)

3. Primary Outcome: Exposure Biomarkers: CEMA
Description: CEMA level after switching to SREC as percentage of baseline level
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of baseline level
Arm/Group | Switching From Smoking Cigarettes to SREC
Number analyzed (Participants) | 23
Percentage of baseline level | 15.0 (20.2)

4. Primary Outcome: Exposure Biomarkers: 3-HPMA
Description: 3-HPMA level after switching to SREC as percentage of baseline level
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: Percentage of baseline level
Arm/Group | Switching From Smoking Cigarettes to SREC
Number analyzed (Participants) | 23
Percentage of baseline level | 38.5 (35.7)

5. Primary Outcome: Inflammatory Biomarkers
Description: Urinary isoprostane level after switching to SREC as percentage of baseline level
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of baseline level
Arm/Group | Switching From Smoking Cigarettes to SREC
Number analyzed (Participants) | 23
Percentage of baseline level | 88.3 (52.6)

6. Primary Outcome: Salivary Biomarkers
Description: Levels of NNN in saliva after switching to SREC
Time Frame: 6 weeks
Population: Only 11 subjects analyzed. Remaining subjects did not have sufficient sample volume for specific analysis.
Measure: Mean (Standard Deviation); unit: pg/mL Saliva
Arm/Group | Switching From Smoking Cigarettes to SREC
Number analyzed (Participants) | 11
pg/mL Saliva | 229.7 (640)

7. Secondary Outcome: Product Use
Description: For cigarettes, cigarettes per day will be assessed based on Interactive Voice Response (IVR) system.
Time Frame: 1 Year
Reporting Status: Not Posted

8. Secondary Outcome: Cigarette Avoidance
Description: The number of cigarette avoidance days, defined as no tobacco cigarettes smoked in the past 24 hours based on IVR, and the rate of cigarette avoidance, calculated as the proportion of cigarette avoidance days out of the total number of days in the product use period (56 days for those who complete the study).
Time Frame: 1 Year
Reporting Status: Not Posted

9. Secondary Outcome: Exposure Biomarkers: Total NNN
Description: Urinary total NNN level (TSNA biomarker) after switching to SREC as percentage of baseline level
Time Frame: 1 Year
Reporting Status: Not Posted

10. Secondary Outcome: Exposure Biomarkers: 1-HOP
Description: Urinary level of 1-HOP (PAH biomarker) after switching to SREC as percentage of baseline level
Time Frame: 1 Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Switching From Smoking Cigarettes to SREC
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 5/47
Other Adverse Events (participants affected / at risk) | 28/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switching From Smoking Cigarettes to SREC (N=47)
Thromboembolic event (DVT/pulmonary embolism) (Vascular disorders) | 1 (1)
Cancer, Lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Head Injury - Accident (Injury, poisoning and procedural complications) | 1 (1)
Pneumonitis (pneumonia) (Infections and infestations) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switching From Smoking Cigarettes to SREC (N=47)
Chest Pain - Cardiac / Angina (Cardiac disorders) | 2 (2)
Tachycardia / Fast heart rate (Cardiac disorders) | 1 (1)
Eye Pain (incl: dry/irritation/itchy/watery) (Eye disorders) | 1 (1)
Periodontal Problem (Gums) (Investigations) | 1 (2)
Vomiting (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Diarrhea (General disorders) | 2 (2)
Tooth Loss (General disorders) | 1 (1)
Cold/clammy/pale skin (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vivid Dreams (see S for nightmare/terror) (General disorders) | 1 (1)
Bronchial Infection (Infections and infestations) | 1 (1)
COVID-19 (Tested + or presumed dx by PCP) (Infections and infestations) | 2 (2)
Fracture (Metabolism and nutrition disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign Cyst/Mass/Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness/Lightheadedness (Investigations) | 2 (2)
Headache (incl. migraine) (General disorders) | 4 (7)
Depressed (sad) mood (General disorders) | 7 (7)
Allergic rhinitis (incl. seasonal allergies) (Immune system disorders) | 4 (4)
Cough (Investigations) | 10 (11)
Nasal congestion (incl. runny nose) (General disorders) | 4 (4)
Nosebleed / Dry nasal membrane (General disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Stress (General disorders) | 1 (1)
Hypertension / Elevated BP (Cardiac disorders) | 3 (3)
Hypotension / Low BP (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT04003805/Prot_SAP_000.pdf